CLINICAL TRIAL: NCT05670795
Title: Comparison of Recombinant Follicle Stimulating Hormone and the Combination of Recombinant Follicle Stimulating Hormone With Clomiphene Citrate in Stimulated Intrauterine Insemination Cycles: A Prospective Randomized Controlled Multicentric Study
Brief Title: Comparison of Recombinant Follicle Stimulating Hormone and the Combination of Recombinant Follicle Stimulating Hormone With Clomiphene Citrate in Stimulated Intrauterine Insemination Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 07.12.2022-E.87948
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Infertility Unexplained
Keywords: ovulation induction; iui
MeSH Terms: interventions — Glycoprotein Hormones, alpha Subunit; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- recombinant follicle stimulating hormone (Experimental): Gonal-f® (75 I.U., Merck Serono, Darmstadt, Germany)
  Interventions: Drug: Recombinant Follicle Stimulating Hormone
- recombinant follicle stimulating hormone and clomiphene citrate (Active Comparator): Gonal-f® (75 I.U., Merck Serono, Darmstadt, Germany) Klomen® (50 mg, Koçak Farma, Tekirdag, Turkey)
  Interventions: Drug: Recombinant Follicle Stimulating Hormone and Clomiphene Citrate

INTERVENTIONS:
Drug: Recombinant Follicle Stimulating Hormone — clinical pregnancy rates
  Arms: recombinant follicle stimulating hormone
Drug: Recombinant Follicle Stimulating Hormone and Clomiphene Citrate — clinical pregnancy rates
  Arms: recombinant follicle stimulating hormone and clomiphene citrate

SUMMARY:
The aim of study is to evaluate the results of two different protocols for ovulation induction during IUI cycles. All patients undergo IUI cycles are randomly divided in to two groups. the first group is recombinant follicle stimulating hormone and the second group is the combination of recombinant follicle stimulating hormone with clomiphene citrate.

DETAILED DESCRIPTION:
Approximately %10-15 of couples of reproductive age, have infertility issues. %30-40 male factor, %40-50 female factor, and %20-25 both play a role in infertility etiology. Contributory factors of cases are %30-40 male factors, %40-50 female factors, and %20-25 mixed type. Ovulation induction and intrauterine insemination (IUI) are the main treatments for infertility. IUI is accepted as the most used treatment procedure according to other assisted reproductive techniques because it has lower costs, can be easily applied, and is less invasive. Clomiphene citrate is the most commonly used for ovulation induction, which is cheaper and has a lower incidence of multiple pregnancies. Controlled ovarian hyperstimulation with recombinant follicle stimulating hormone and IUI has a higher incidence of pregnancy rates in an ovulation, unexplained and mild male factor infertility cases.

Data including age, BMI, smoking, the duration of infertility, the type of infertility, total motile sperm count (TMSS) of inseminated material and sperm morphology, antral follicle count, number of developed follicles and endometrial thickness on HCG day will be recorded. On the 2nd or 3rd day of the cycle, the patient will be randomized into two groups. Group 1 (rFSH: n=127, 75 IU FSH/day), and Group 2 (clomiphene citrate 100 mg/day for 5 days following by 75 IU FSH/day; n=127). Human chorionic gonadotropin (hCG) will be used for trigger when the dominant follicle's diameter reaches 17-18mm for ovulation. Thirty-six hours after the hCG injection, single IUI will be performed by using the fresh sperm obtained by the density gradient method with a soft catheter in the dorsolithotomy position under ultrasound guidance. The patient will be kept supine position after the procedure for 15 minutes. After IUI, sexual intercourse will be recommended for three days. Intravaginal progesterone (LUTINUS® 100 mg vaginal tablet, Ferring GmbH Wittland/Kiel/Germany) to both groups will be used once a day after insemination for luteal phase support. Clinical pregnancy rates will be recorded by performing a blood test for on the 15th day after the procedure.

The aim of study is to evaluate the results of two different protocols for ovulation induction during IUI cycles. All patients undergo IUI cycles are randomly divided in to two groups. the first group is recombinant follicle stimulating hormone and the second group is the combination of recombinant follicle stimulating hormone with clomiphene citrate

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old female
* Unexplained infertility
* Regular menstrual cycle
* Bilateral tubal patency in HSG and normal uterine cavity
* Total motile sperm count greater than 10 million/ml

Exclusion Criteria:

* History of ovarian surgery
* Uncorrected uterine pathology
* Other endocrine diseases (thyroid, prolactin, hypogonadotropic hypogonadism)
* Presence of a cyst greater than 10 mm on USG in 2-3 days of the period
* Stage 3-4 endometriosis
* TMSS < 5 million/ml on the insemination day
* Conditions where rFSH and clomiphene citrate are contraindicated

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 254 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical pregnancy | day 15
  after iui betahcg levels blood sampling

SECONDARY OUTCOMES:
Rate of ongoing pregnancy | Months 3
  Ongoing pregnancy rates 3 months after iui

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peeraer K, Debrock S, De Loecker P, Tomassetti C, Laenen A, Welkenhuysen M, Meeuwis L, Pelckmans S, Mol BW, Spiessens C, De Neubourg D, D'Hooghe TM. Low-dose human menopausal gonadotrophin versus clomiphene citrate in subfertile couples treated with intrauterine insemination: a randomized controlled trial. Hum Reprod. 2015 May;30(5):1079-88. doi: 10.1093/humrep/dev062. Epub 2015 Mar 18. PMID 25788569
- [Background] Erdem M, Abay S, Erdem A, Firat Mutlu M, Nas E, Mutlu I, Oktem M. Recombinant FSH increases live birth rates as compared to clomiphene citrate in intrauterine insemination cycles in couples with subfertility: a prospective randomized study. Eur J Obstet Gynecol Reprod Biol. 2015 Jun;189:33-7. doi: 10.1016/j.ejogrb.2015.03.023. Epub 2015 Mar 28. PMID 25855325
- [Background] Dankert T, Kremer JA, Cohlen BJ, Hamilton CJ, Pasker-de Jong PC, Straatman H, van Dop PA. A randomized clinical trial of clomiphene citrate versus low dose recombinant FSH for ovarian hyperstimulation in intrauterine insemination cycles for unexplained and male subfertility. Hum Reprod. 2007 Mar;22(3):792-7. doi: 10.1093/humrep/del441. Epub 2006 Nov 16. PMID 17110396